CLINICAL TRIAL: NCT04289350
Title: Day to Day Variation in Fetal Heart Rate Variability Based on Fetal Electrocardiography (FECG), in a Standardized Setting: A Cohort Study
Brief Title: Day to Day Variation in Fetal Heart Rate Variability
Acronym: (FHRV)
Status: Completed | Type: Observational
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other); Snedkermester Sophus Jacobsen and hustru Astrid Jacobsens Foundation (Other); Hartmann Fonden (Other); Augustinus Fonden (Other); The Dagmar Marshall Foundation (Other); AP Moeller Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: fHRV_2
Record Dates: First submitted 2020-02-20; First posted 2020-02-28 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2020-02

CONDITIONS: Fetal Growth Retardation
MeSH Terms: conditions — Fetal Growth Retardation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Diagnostic Test: fetal heart rate variability — An observational study. No intervention

SUMMARY:
This study evaluates the day-to-day variation in fetal heart rate variability based on non-invasive fetal-ECG (NI-FECG). Furthermore, the effect of fetal movements on fetal heart rate variability will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Healthy singleton pregnant women with an expected healthy fetus

Exclusion Criteria:

* fetal malformations, multiple pregnancy, obstetric complications, maternal chronic disease and labor. Low birth weight or malformation diagnosed at birth.

Sex: Female
Age Groups: Child, Adult, Older Adult
Study Population: Healthy singleton pregnant women. Danish.
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Root mean square of successive inter beat interval differences (RMSSD) | 1/8-2020
  Time domain analysis
Standard deviation of normal to normal inter beat interval (SDNN) | 1/8-2020
  Time domain analysis
High frequency power (HF-power) | 1/8-2020
  Spectral analysis
Low frequency power (LF-power) | 1/8-2020
  spectral analysis
Low frequency power/High frequency power (LF/HF) | 1/8-2020
  Spectral analysis

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Obstetrics and Gynecology. Aarhus Unive, Aarhus, Aarhus N, Denmark

IPD SHARING:
Plan to Share IPD: No